CLINICAL TRIAL: NCT00704236
Title: Phase 4 Study on the Effect of Insulin Resistance With Traditional Chinese Treatment in Type 2 Diabetes
Brief Title: Improvement of Insulin Resistance With Traditional Chinese Treatment in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCEMD003
Record Dates: First submitted 2008-06-16; First posted 2008-06-24 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Type 2 Diabetes
Keywords: Traditional Chinese Treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Coptidis rhizoma extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Coptis Chinensis, Astragalus mambranesceus, Lonicera Japonica (Traditional Chinese Treatment)
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coptis Chinensis, Astragalus mambranesceus, Lonicera Japonica (Traditional Chinese Treatment) — 50 mg of Coptis Chinensis, 30 mg of Astragalus mambranesceus and 120 mg of Lonicera Japonica
  Arms: A
Drug: Placebo
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the efficacy of Traditional Chinese Treatment(TCT) on insulin sensitivity and other related factors in type 2 diabetes by using an double-blind, randomized, parallel control and prospective study This traditional compound Chinese herb preparation is referred to this study, with three kinds of plants: 50 mg of Coptis Chinensis, 30 mg of Astragalus mambranesceus and 120 mg of Lonicera Japonica, all of which are selected by The Chinese Academy of Medical Sciences among those traditionally considered effective and safe in the treatment of diabetes.

Patients enrolled were randomized into TCT group and placebo group administrated with TCT and placebo respectively. Glucose disposal rate (GDR), fasting plasma glucose (FPG), postprandial plasma glucose (PPG), HbA1C and other metabolic components were assessed at baseline and end point

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed type 2 diabetes poorly controlled by diet only for one month
2. Obese with a BMI of 23-35 kg/m2

Exclusion Criteria:

1. Those patients used any drugs for treatment of diabetes
2. Patients with evidence of cardiac, hepatic, renal, other chronic diseases or acute diabetic complications including diabetic ketoacidosis or hyperosmolar hyperglycemic non-ketotic coma
3. Women who were pregnant or planned pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-09; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Glucose Disposal Rate

SECONDARY OUTCOMES:
Fasting Plasma Glucose,Postprandial Plasma Glucose,HbA1c,triglyceride,cholesterol,HDL-c and LDL-c,lipid levels ,body weight, blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD. PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China